CLINICAL TRIAL: NCT02367625
Title: Performance, Safety, and Efficacy of a New Cyrotherapy Device for Cervical Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1UH2CA189923-01 (NIH)
Record Dates: First submitted 2014-12-27; First posted 2015-02-20 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): 20 women with normal cervical cytology will be randomized to receive MedGYn MGC 200 therapy
  Interventions: Device: CryoPop
- Arm 2 (Active Comparator): 20 women with normal cervical cytology will be randomized to receive MedGYn MGC 200 therapy
  Interventions: Device: MedGyn MGC 200

INTERVENTIONS:
Device: CryoPop — The new CryoPop device will be compared to standard cryotherapy
  Arms: Arm 1
Device: MedGyn MGC 200 — Standard cryotherapy
  Arms: Arm 2

SUMMARY:
Globally, cervical cancer is the second most common cancer for women and kills approximately 250,000 women every year, with the annual number of deaths expected to increase to 410,000 by 2030. The majority (88%) of these deaths occur in low- and middle-income countries (LMICs) where screening and prevention services are limited. Prevention of cervical cancer by identification and treatment of cervical cancer precursors is key, since treatment resources for invasive disease are scarce. A cervical cancer screening program cannot be effective unless it is linked with a proven intervention to prevent the development of cervical cancer. The World Health Organization (WHO) recently released the WHO guidelines for screening and treatment of precancerous lesions for cervical cancer prevention, which recommends a screen-and-treat approach for cervical cancer prevention, with cryotherapy being the first choice of treatment for women who have a positive screen. However, these programs are still slow to be implemented in part due to the current high cost and low efficiency of cryotherapy equipment that is often prone to breaking. Jhpiego, an affiliate of Johns Hopkins University, has developed a new cryotherapy device, CryoPop, that is one tenth the cost of current equipment while also ten times more efficient. Once proven safe, feasible and effective, CryoPop could save tens of thousands of lives in low- and middle-income countries each year by preventing cervical cancer.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recently released the WHO guidelines for screening and treatment of precancerous lesions for cervical cancer prevention23 which recommends a screenand- treat approach for cervical cancer prevention (CECAP), with cryotherapy being the first choice of treatment for women who have a positive screen. Cryotherapy using nitrous oxide (N2O) or carbon dioxide (CO2) to induce cryonecrosis of dysplastic tissues followed by regeneration of normal cervical epithelium is the most common intervention used in LMICs because it is simple and safe enough for mid-level providers such as nurses or midwives to operate, and can be performed without anesthesia or electricity.

CO2 is more often used than N2O due to its wider availability and lower cost. Mid-level providers have been trained successfully to perform cryotherapy safely and with a high degree of acceptability.24,25,26 Adverse effects after cryotherapy are relatively uncommon and generally minor, reported in 1-2% of women. A recent meta-analysis of the effectiveness of cryotherapy found cure rates of 85% and 92%, respectively, in CIN 2 and CIN 3. An alternative to cryotherapy, loop electrosurgical excisional procedure (LEEP) has largely supplanted cryotherapy in well-resourced settings, as it provides a surgical specimen for pathologic assessment and can be used on large lesions ineligible for cryotherapy. However, LEEP requires electricity, is more costly, requires a higher level of training and is associated with a higher rate of complications, all of which complicate its routine use in LMICs. While LEEP may be available in national referral centers, WHO recommends cryotherapy in settings where it is not available. Cost, reliability, durability and reparability are all factors that prohibit the scale-up necessary for current cryotherapy methods to match the volume of population-based screening needed to achieve a marked decrease in cervical cancer morbidity and mortality. Each cryotherapy unit costs approximately $2,000, resulting in approximately 80% of the treatment cost of cryotherapy being directly attributed to equipment cost. Additionally, the design involves many custom parts available only through the manufacturers, which are all based in the U.S. or Europe. This prohibits local repairs and limits the life of the product to only one or two years (or even less when spare parts are not available). Cryoguns were initially developed for use with N2O but they can be used with CO2. CO2 is approximately one fifth of the cost of N2O; however CO2, in its various usage, from recreational to medical grade, is less regulated and often of variable purity and concentration-leading to more equipment failures. Last but not least, the design of the equipment makes it inefficient with the use of CO2 gas, increasing cost and missed opportunities while the gas cylinder is being refilled at a central gas supply depot. In most LMICs, this means sending the gas cylinder to the capital city. On average, a single 50lb CO2 tank can treat only 10 to 15 women. The subject of this proposal, CryoPop, is a new technology specifically designed for LMIC settings and more appropriate to support see-and-treat efforts because of its low cost and durability. The CryoPop device is currently expected to cost one tenth of the price of current devices while also using one tenth of the CO2 supply, thereby substantially reducing purchase price coupled with far greater efficiency in the use of CO2, making the CryoPop attractive for further investment. Moreover, this device is designed to have minimum moving components which at the same time are inexpensive to replace and easy to repair in-situ by the providers themselves. Finally, the CryoPop is not tethered to the gas canister during the procedure, adding more safely to the process by not having to be concerned over tank or gas line placement. The goal is to have a device for the frontline where screening is happening and provide the unique opportunity of minimizing if not preventing loss to follow-up of screen-positive women.

This will accelerate access to cervical cancer prevention and treatment services by enabling implementation of SVA to rural, underdeveloped regions, most of which have never had CECAP programs.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 30-49 years old
2. Must have normal cervical cytology
3. Must have planned total hysterectomy for other gynecological indication

Exclusion Criteria:

1. Menopause
2. Past history of cervical dysplasia
3. Known HIV+or history of other sexually transmitted infections -

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
The primary variable of interest is the width of necrosis on the cervical pathologic specimen | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jean Anderson, MD, Study Director — Jhpiego
Locations (1):
- University of the Phillipines, College of Medicine, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Undecided